CLINICAL TRIAL: NCT00643071
Title: Tacrolimus (FK506) P-III, Open-label Study in Severe Refractory Ulcerative Colitis Patients or Patients Who Attended and Received Placebo in F506-CL-1107 Study
Brief Title: Tacrolimus (FK506) P-III, Open-label Study in Refractory Ulcerative Colitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F506-CL-1108
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Tacrolimus; FK506; Treatment outcome
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Oral
  Other Names: FK506

SUMMARY:
Patients with severe refractory ulcerative colitis (UC) or those who received placebo in study F506-CL-1107 will receive tacrolimus for a maximum of 12 weeks. Safety and efficacy will be evaluated.

DETAILED DESCRIPTION:
Patients with severe refractory ulcerative colitis (UC) or those who received placebo in study F506-CL-1107 study can participate in this study. Patients will receive tacrolimus for a maximum of 12 weeks in an open-label study manner. Improvement of Disease Activity Index (DAI) score and other efficacy scores will be evaluated during the drug administration period.

ELIGIBILITY:
Inclusion Criteria:

* Severe refractory UC patients who meets the following criteria

  * Disease activity: more than 6 times of stool a day, bloody stool, moderate to severe endoscopic finding
  * Steroid resistant or dependent

OR

* Moderate to severe refractory UC patients who participated and received placebo in F506-CL-1107 study

Exclusion Criteria:

* Mild or fulminant type
* Renal failure patients, hepatic failure patients
* Patients taking 6-mercaptopurine, cyclosporin or other immunosuppressants within 12 weeks prior to entry
* Patients who received LCAP or GCAP within 2 weeks prior to entry
* Patients who changed the dose of steroid or started steroid within 2 weeks prior to entry
* Patients who changed the dose of steroid or started steroid within 1 week prior to entry in case they received more than 40 mg/ day or 1mg/kg/day of steroid just before the study

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Improvement of Disease Activity Index score (DAI score) | 12 weeks

SECONDARY OUTCOMES:
Changes of DAI score ( Total & each item) | 2 weeks
Changes of clinical severity and symptom | 12 weeks
Endoscopic finding | 12 weeks
Patients impression | 12 weeks
Amount of steroid | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu
  - Shin'etsu